CLINICAL TRIAL: NCT04449523
Title: Incidence of Silent Atrial Fibrillation in Patients With Clinically Silent Brain Ischemic Lesions (SILENT2)
Brief Title: Incidence of Silent Atrial Fibrillation in Patients With Clinically Silent Brain Ischemic Lesions
Acronym: SILENT2
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-00227
Record Dates: First submitted 2020-06-17; First posted 2020-06-29 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Silent Stroke; Silent Cerebral Infarct; Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Arterial Fibrillation (AF) is well-recognized as a cause for cryptogenic Acute Ischemic Stroke (AIS) and is associated with Silent Brain Infarction (SBI). However, the role of AF in the formation of lesions (SBIs) is less well established than its role in AIS and needs clarification.

The investigators hypothesize that continuous rhythm monitoring will yield a similar incidence of AF diagnosis in patients with SBI as compared to patients with cryptogenic AIS.

The primary objective is to assess the cumulative incidence of AF diagnosis at 24 months in patients with SBI.

DETAILED DESCRIPTION:
Arterial Fibrillation (AF) is well-recognized as a cause for cryptogenic Acute Ischemic Stroke (AIS) and searched for in clinical practice. However, although AF is associated with Silent Brain Infarction (SBI), its role in the formation of these lesions is less well established and needs clarification. A multitude of clinical, laboratory, echocardiographic and electrocardiographic parameters are associated with AF. Although no single one of these parameters has sufficient specificity to rule-in AF, their combined use may nevertheless help to identify patients with SBI at highest risk for AF. The study is expected to provide evidence that long term monitoring in subjects with SBI yields similar rates of AF as in AIS patients.

Patients aged ≥65 years with a presumably silent brain lesion in a brain magnetic resonance imaging fulfilling inclusion criteria and consenting get a subcutaneous implantation of a cardiac monitor (Reveal LINQ). Data will be directly transferred to the treating physician by the Medtronic MyCareLink Patient Monitor. In case of a relevant arrhythmia, the respective study site will be informed by the staff of Inselspital. Relevant arrhythmias are defined as follows:

* First episode of atrial fibrillation (≥30 seconds)
* Sustained ventricular tachycardia (≥30 seconds)
* Sustained supraventricular tachycardia (≥30 seconds)
* Asystoly of ≥6 seconds duration
* Atrial fibrillation with pause of ≥6 seconds duration
* Higher degree atrioventricular (AV) block (3° AV bloc; 2:1 AV conduction; 2° AV block type Mobitz)
* Sustained bradycardia <30 beats per minute (≥30 seconds) It is the responsibility of the respective study sites to take appropriate actions and inform the patients and treating physicians about relevant findings. The maximal timeframe from data transmission to data analysis is one week and from data transmission to patient notification two weeks.

The expected results of the study would be supportive in introducing long term monitoring to the care pathway in subjects with SBI. Since SBI are more prevalent than AIS and current recommendations very restrictive, this would have a relevant impact on SBI management.

ELIGIBILITY:
Inclusion Criteria:

* Age

  * ≥ 65 years
  * ≥ 50 years AND one the following:

    * NT-proBNP >400 pg/mL
    * Left atrial ventricular index >42 ml/m2 or left atrial diameter >46 mm
    * Covert infarctions with cortical involvement in more than one vascular territory (left carotid territory, right carotid territory, vertebrobasilar territory)
* Written informed Consent
* Any clinically silent ischemic lesions of the brain parenchyma detected on neuroimaging defined according to established criteria as either:

  * Diffusion weighted imaging (DWI) positive lesions: Focus of restricted diffusion (high DWI signal and low apparent diffusion coefficient value) occurring in either white or gray matter, located in the cerebrum, cerebellum, or brain stem AND not satisfying the diagnostic criteria for multiple sclerosis OR
  * Cavitatory Lesions: ≥ 3 mm in size that follow cerebro-spinal fluid on all sequences that are slit or wedge shaped with an irregular margin AND NOT longitudinally aligned with perforating vessels or with a multiple, bilateral symmetrical distribution OR
  * T2 weighted (T2W) hyperintense/T1 weighted (T1W) hypointense lesions:

    * Focal lesion with high T2W signal and low T1W signal that have prior evidence of restricted diffusion; OR
    * Present within cortical gray matter or deep gray matter nuclei OR
    * A lesion that is new, compared with an MRI performed within 3 months OR
    * T2W hyper/T1W hypointense lesions in the white matter, which are discontinuous but associated with the classic confluent periventricular T2 intense change of leukoaraiosis (Fazekas ≥2) AND NOT satisfying the diagnostic criteria for multiple sclerosis or with a significant patient history of severe trauma, radiation, drug toxicity, or carbon monoxide poisoning

Exclusion Criteria:

* History of AF or atrial flutter
* Patients with a history of symptoms compatible with an AIS, covert neurological deficits are allowed.
* Cardiac implantable electronic devices (pacemaker, implantable cardiac defibrillator (ICD), implantable cardiac monitor (ICM))
* Indication for cardiac implantable electronic device implantation (pacemaker, ICD, ICM)
* History of or indication for major cardiac surgery or transcutaneous aortic valve implantation
* Indication for permanent oral anticoagulation
* Contraindication for permanent oral anticoagulation
* Projected life expectancy of less than 2 years
* Active intra- or extracranial high-grade malignancy
* Patient is already included in another clinical trial that will affect the objectives of this study
* Patient's lack of accountability, inability to appreciate the nature, meaning and consequences of the study and to formulate his/her own wishes correspondingly
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.
* Known or suspected non-compliance, drug or alcohol abuse

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ≥ 50 years
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-09-08 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of Arterial Fibrillation (AF) diagnosis over a median of 24 months | From day 0 to 24 months after inclusion
  Only adjudicated events will be used for the analysis. An AF episode is defined as lasting more than 30 seconds. A diagnosis of atrial flutter will also be considered as a primary endpoint.

SECONDARY OUTCOMES:
Time to first diagnosis of AF (lasting ≥30 seconds; ≥6 minutes; ≥1 hour; ≥ 24 hour) | From day 0 to 24 months after inclusion
Burden of AF | From day 0 to 24 months after inclusion
  The burden of AF is defined as the amount of time (percentage) in AF during rhythm monitoring. AF burden will be calculated on a monthly basis.
Time to composite of first diagnosis of AF, stroke and death. | From day 0 to 24 months after inclusion
Incidence of AF diagnosis according to Silent Brain Infarction (SBI) neuroradiological appearance (subcortical small vessel versus embolic pattern involving grey matter) and SBI fulfilling ESUS criteria versus lacunar type. | From day 0 to 24 months after inclusion
  Embolic stroke of undetermined source (ESUS)
Start of oral anticoagulation therapy at 24 months. | At 24 months
Stroke at 24 months | At 24 months
Mortality at 24 months | At 24 months
Prevalence of other possible etiologies for SBI according to a modified TOAST-classification (large artery disease, small artery disease, other specific etiologies, unknown etiology, incomplete workup) | From day 0 to 24 months after inclusion
Incidence of new SBI at 24 months (only if sufficient funding can be obtained for repeat brain MRI at 24 months without contrast agent) | At 24 months

OTHER OUTCOMES:
Time to first diagnosis of AF (lasting ≥30 seconds; ≥6 minutes; ≥1 hour; ≥ 24 hours) until battery depletion of Implantable Cardiac Monitor (ICM) (36-42 month). | From day 0 until battery depletion, expected to be 36 to 42 months
Cumulative incidence of AF diagnosis until battery depletion of ICM | From day 0 to until battery depletion, expected to be 36 to 42 months

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Roten, PD Dr. med., Principal Investigator — Inselgruppe AG
Locations (8):
- Universitätsspital Graz, Graz, Austria
- Charite Berlin, Berlin, Germany
- Switzerland (6):
  - Centre hospitalier universitaire vaudois (CHUV), Lausanne, Canton of Vaud
  - Kantonsspital Aarau, Aarau
  - University Hospital Basel, Basel
  - Inselspital Bern, Bern
  - Kantonsspital St.Gallen, Sankt Gallen
  - Universitätsspital Zurich, Zurich